CLINICAL TRIAL: NCT07049068
Title: Double-bllind, Double-dummy, Randomized Clinical Trial Comparative Between Oral Nicotinamide Versus Topical Nicotinamide in the Management of Facial Actinic Keratosis .
Brief Title: Comparison of Nicotinamide Treatments for Actinic Keratosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Univates (Other)
Responsible Party: Principal Investigator, Thais Cachafeiro, Principal investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 52100621.0.0000.5347
Record Dates: First submitted 2025-06-07; First posted 2025-07-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Actinic Keratoses
Keywords: actinic keratosis; nicotinamide; topical nicotinamide; oral nicotinamide
MeSH Terms: conditions — Keratosis, Actinic | interventions — Niacinamide

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, double-dummy clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral nicotinamide (group 1) (Active Comparator): Received 120 capsules of 500 mg nicotinamide and a tube of placebo cream at each visit.
  Interventions: Drug: Oral Nicotinamide
- topical nicotinamide (group 2) (Active Comparator): Participants from group 2 received a tube of 5% nicotinamide cream and 120 placebo capsules.
  Interventions: Drug: topical nicotinamide

INTERVENTIONS:
Drug: Oral Nicotinamide — Participants from group 1 received 120 capsules of 500 mg nicotinamide and a tube of placebo cream at each visit. . All participants were instructed to take 1 capsule every 12 hours and to apply the cream to their entire face twice a day.
  Participants were unaware of which group they were allocated to and participants in both groups received either capsules (active or placebo, which looked identical) or a tube of cream (active or placebo, which looked identical). In follow-up visits participants returned empty tubes to the responsible pharmacist.
  At the initial assessment and at 6 months photographs of the participants' faces were taken.
  Arms: oral nicotinamide (group 1)
Drug: topical nicotinamide — Participants from group 2 received a tube of 5% nicotinamide cream and 120 placebo capsules. All participants were instructed to take 1 capsule every 12 hours and to apply the cream to their entire face twice a day.
  Participants were unaware of which group they were allocated to and participants in both groups received either capsules (active or placebo, which looked identical) or a tube of cream (active or placebo, which looked identical). In follow-up visits participants returned empty tubes to the responsible pharmacist.
  At the initial assessment and at 6 months photographs of the participants' faces were taken.
  Arms: topical nicotinamide (group 2)

SUMMARY:
In this study, the investigators aimed to evaluate the effect of oral nicotinamide compared to topical nicotinamide in the presence of actinic keratoses on the face. The reason that led the investigators to study this subject is that previous studies have shown possible favorable effects of nicotinamide, both topical and oral, in the prevention of precursor lesions of skin cancer. However, there are no studies to date comparing topical and oral presentations of nicotinamide in the prevention of the appearance of actinic keratoses and in the regression of the number of actinic keratoses.

In this randomized clinical trial, 74 participants with actinic keratoses on the face received either oral nicotinamide and topical placebo or topical nicotinamide and oral placebo for 6 months.

DETAILED DESCRIPTION:
Background: Nicotinamide has been reported to be effective in reducing rates of actinic keratosis, however, to date, there are no studies comparing their topical and oral presentations Objectives: to compare efficacy of oral and topical nicotinamide in preventing and reducing the number of facial actinic keratosis. Secundary objectives: to evaluate the occurrence of non-melanoma skin cancer (NMSC) and evaluate the safety and adverse effect profile of topical and oral nicotinamide.

Methods: In this randomized, double-blind, double-dummy clinical trial, 74 participants with actinic keratosis on the face received either oral nicotinamide and topical placebo or topical nicotinamide and oral placebo for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* male individuals over 18 years of age
* female individuals with tubal ligation, hysterectomy or over 45 years of age in menopause
* presence of at least three palpable actinic keratoses on the face

Exclusion Criteria:

* individuals with an incidence of 3 or more squamous cell carcinomas in the last year
* solid organ transplant recipients
* carriers of the human immunodeficiency virus (HIV)
* solid organs cancer
* active gastric ulcer
* recent history of acute myocardial infarction
* hypotension
* pregnancy
* lactation
* chronic liver disease
* liver or kidney failure
* xeroderma pigmentosum
* albinism
* epidermodysplasia verruciformis
* dystrophic epidermolysis bullosa
* nevoid basal cell carcinoma syndrome
* individuals with a large number of confluent actinic keratosis (making it impossible to count individual lesions)
* Individuals using carbamazepine
* Individuals using oral retinoids
* Individuals using oral supplements containing nicotinamide
* Individuals who had undergone field treatments for actinic keratoses such as 5-fluorouracil in the last 4 months
* individuals who were unable to understand the objectives and risks of treatment
* Individuals who refused to participate or sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
facial actinic keratosis in 6 months | From enrollment to the end of treatment at 6 months
  The primary outcome is the number of facial actinic keratosis after 6 months of treatment (compared with baseline).

SECONDARY OUTCOMES:
facial actinic keratosis in 2 months | From enrollment to the 2 months treatment
  number of actinic keratosis on the face after 2 months of treatment (compared with baseline)
facial actinic keratosis in 4 months | From enrollment to 4 months treatment
  number of actinic keratosis on the face after 4 months of treatment (compared with baseline)
number of squamous cell carcinomas and basal cell carcinomas after 2 months | from baseline to 2 months treatment
  number of squamous cell carcinomas and basal cell carcinomas in the treated area and on the whole body after 2 months of treatment (compared with baseline).
number of squamous cell carcinomas and basal cell carcinomas after 4 months | from enrollment to 4 months treatment
  number of squamous cell carcinomas and basal cell carcinomas in the treated area and on the whole body after 4 months
number of squamous cell carcinomas and basal cell carcinomas after 6 months | from enrollment to 6 months treatment
  number of squamous cell carcinomas and basal cell carcinomas in the treated area and on the whole body after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Programa de Pós Graduação Ciencias Médicas UFRGS, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
sex, age, number of actinic keratosis
Supporting Information: Study Protocol, CSR
Time Frame: from now for 3 years

REFERENCES:
- [Background] Surjana D, Halliday GM, Martin AJ, Moloney FJ, Damian DL. Oral nicotinamide reduces actinic keratoses in phase II double-blinded randomized controlled trials. J Invest Dermatol. 2012 May;132(5):1497-500. doi: 10.1038/jid.2011.459. Epub 2012 Feb 2. No abstract available. PMID 22297641
- [Background] Moloney F, Vestergaard M, Radojkovic B, Damian D. Randomized, double-blinded, placebo controlled study to assess the effect of topical 1% nicotinamide on actinic keratoses. Br J Dermatol. 2010 May;162(5):1138-9. doi: 10.1111/j.1365-2133.2010.09659.x. Epub 2010 Mar 1. No abstract available. PMID 20199551
- [Background] Sivapirabu G, Yiasemides E, Halliday GM, Park J, Damian DL. Topical nicotinamide modulates cellular energy metabolism and provides broad-spectrum protection against ultraviolet radiation-induced immunosuppression in humans. Br J Dermatol. 2009 Dec;161(6):1357-64. doi: 10.1111/j.1365-2133.2009.09244.x. Epub 2009 Apr 20. PMID 19804594
- [Background] Chen AC, Martin AJ, Choy B, Fernandez-Penas P, Dalziell RA, McKenzie CA, Scolyer RA, Dhillon HM, Vardy JL, Kricker A, St George G, Chinniah N, Halliday GM, Damian DL. A Phase 3 Randomized Trial of Nicotinamide for Skin-Cancer Chemoprevention. N Engl J Med. 2015 Oct 22;373(17):1618-26. doi: 10.1056/NEJMoa1506197. PMID 26488693

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT07049068/Prot_SAP_000.pdf